CLINICAL TRIAL: NCT03206229
Title: A Randomized, Double Blind, Single-Dose, Two-Period Crossover Comparative Pharmacology Study Comparing TPI-120 and Neulasta® Administered Through Subcutaneous Route in Healthy Adult Subjects
Brief Title: Study Comparing TPI-120 and Neulasta Administered Through Subcutaneous Route in Healthy Adult Subjects
Acronym: TPI-120
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adello Biologics, LLC (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Principal Investigator, Dr. Apinya Vutikullid, principal investigator, Adello Biologics, LLC
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TPI-CL-109-A
Record Dates: First submitted 2017-04-12; First posted 2017-07-02 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor; pegfilgrastim

STUDY DESIGN:
Intervention Model Description: This study is a Randomized, Double Blind, Single-Dose, Two-Period Crossover Comparative Pharmacology Study
Who Masked: Participant, Investigator
Masking Description: This is double blind study so participat healthy subjects and investigators both would be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPI-120 (PEG-rhG-CSF) (Experimental): PEG-rhG-CSF (recombinant granulocyte-colony stimulating factor conjugated with monomethoxypolyethylene glycol) Adello Biologics, LLC, Chicago, IL
  Interventions: Drug: PEG-rhG-CSF
- Neulasta (PEG-rhG-CSF) (Active Comparator): Neulasta®, (PEG-rhG-CSF) Amgen, Thousand Oaks, CA
  Interventions: Drug: Neulasta (PEG-rhG-CSF)

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF is going to be administered 2 mg/0.2 ml subcutaneously single dose in each study period as per the randomization schedule
  Other Names: PEGFILGRASTIM
  Arms: TPI-120 (PEG-rhG-CSF)
Drug: Neulasta (PEG-rhG-CSF) — PEG-rhG-CSF is going to be administered 2 mg/0.2 ml subcutaneously single dose in each study period as per the randomization schedule
  Other Names: PEGFILGRASTIM
  Arms: Neulasta (PEG-rhG-CSF)

SUMMARY:
This is a single or up to 2 centers, double-blind, randomized, single-dose, two-way, crossover study comparing the Test (T) and Reference (R) products following subcutaneous administration. Subjects will be randomly assigned to one of two treatments sequences (TR or RT).

All subjects will be dosed at the CRO's designated clinical site(s) and the same protocol requirements and procedures will be followed within each group.

DETAILED DESCRIPTION:
The current study design was prepared to assess and compare the PK, PD, safety, tolerability of the Adello biosimilar candidate, TPI-120 and the US-licensed reference product, Neulasta® after administering a single subcutaneous 2 mg dose in healthy adult subjects in a crossover design. The primary PK parameters are AUC0-t, AUC0-inf, and Cmax, and the primary PD parameters are baseline-corrected AUEC0-t and Emax for ANC.

This is a single or up to 2 centers, double-blind, randomized, single-dose, two-way, crossover study comparing the Test (T) and Reference (R) products following subcutaneous administration. Subjects will be randomly assigned to one of two treatments sequences (TR or RT).

All subjects will be dosed at the CRO's designated clinical site(s) and the same protocol requirements and procedures will be followed within each group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to dosing), 19 - 55 years of age (inclusive), with body mass index (BMI) ≥ 19 and ≤ 30 kg/m2, and body weight not < 50 kg or > 100 kg at the time of screening.
2. Healthy as defined by:

   1. The absence of clinically significant (in the opinion of the PI/designee) illness or surgery within 4 weeks prior to dosing.
   2. The absence of a clinically significant (in the opinion of the PI/designee) history of disease.
   3. WBC (white blood cell) > 4.0 x 109/L and < 1.5 times the upper limit of normal (ULN), ANC (absolute neutrophil count) > 2.0 x 109/L and < 1.5 times the upper limit of normal (ULN), Platelet count > 150 x 109/L, AST (aspartate aminotransferase) < 2.5 time the upper limit of normal (ULN), ALT (alanine aminotransferase) < 2.5 time the upper limit of normal (ULN), Serum bilirubin < 1.5 time the upper limit of normal (ULN) and Serum creatinine < 1.5 time the upper limit of normal (ULN). [Refer to APPENDIX 1 for normal reference ranges]
   4. The absence of febrile (defined by a documented oral temperature of 101.5 °F or greater) or infectious illness within 1 week of first dosing.
   5. The absence of a clinically significant history of skin disorders, including psoriasis.
3. Females of childbearing potential must be willing to use acceptable contraceptive methods throughout the study, and for 30 days thereafter.
4. Females of non-childbearing potential must have undergone sterilization procedures, at least 6 months prior to the first dose or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
5. Capable of consent.
6. Male subjects willing to follow approved birth control method for the duration of the study, and for 30 days thereafter, such as (a double barrier method) vasectomy, condom with spermicide, condom with diaphragm or abstinence, subject should also not donate sperm during this time.

Exclusion Criteria:

1. Positive test for hepatitis B, hepatitis C, or HIV.
2. Illicit/illegal drug use as evidenced by a positive test for alcohol or drug screen at screening or check -in.
3. Positive result for urine alcohol test at screening or check-in
4. Tobacco use as evidenced by a positive cotinine result at screening or check-in.
5. History of allergic reactions to pegfilgrastim, filgrastim, Escherichia coli (E. coli)-derived proteins, or other related drugs. History of allergic reactions or hypersensitivity to acetate/acetic acid, polysorbate 20, or sorbitol.
6. Hereditary fructose intolerance.
7. Females with positive pregnancy tests at screening or check-in.
8. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study or completing follow-up activities.
9. Clinically significant ECG or vital sign abnormalities at screening.
10. History of significant alcohol abuse within one year prior to initial dosing or regular use of alcohol (more than 14 units of alcohol per week) within six months prior to initial dosing.
11. History of drug abuse or use of illicit/illegal drugs within 1 year prior to initial dosing.
12. No medications are permitted during the study. Exceptions are:

    1. Hormonal contraceptives and Hormone Replacement Therapy (HRT),
    2. Thyroid replacement therapy i.e., liothyronine (T3) or levothyroxine (T4).
    3. Acetaminophen
13. Donation of plasma within 7 days of dosing; blood donation or significant loss of blood within 30 days of dosing.
14. Participation in a clinical trial involving the administration of an investigational drug or marketed drug within 30 days prior to initial dosing (90 days for biologics) or concomitant participation in an investigational study involving no drug administration.
15. Females who are breast-feeding or lactating.
16. History of pulmonary infiltrate or pneumonia (radiologically confirmed) within 6 months prior to initial dosing.
17. Any past exposure to recombinant human G-CSF products and/or a known history of prior treatment with blood-cell colony stimulating factors, interleukins or interferons.
18. History of cancer
19. Subjects who are on a special diet or who have self-reported a weight loss of more than 15 pounds within 1 month prior to initial dosing.
20. Acute viral or bacterial infection within 1 month prior to initial dosing only if considered clinically significant in the opinion of the Principal Investigator/designee.
21. History of any clinically significant disease or condition that, in the opinion of the Principal Investigator/designee, would render them unsuitable for inclusion in the study.
22. Any vaccination (including influenza) within 90 days prior to initial dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | 56 days
  To evaluate the pharmacokinetics
Area under the concentration-time curve from time zero to the time of the last non-zero concentration (AUC0-t) | 56 days
  To evaluate the pharmacokinetics
Area under the concentration-time curve from time zero to infinity (extrapolated AUC0-inf) | 56 days
  To evaluate the pharmacokinetics

SECONDARY OUTCOMES:
Safety Variable - Tolerability as measured by Injection Site reactions | 1, 2, 4, and 24 hours postdose during each study period
  Tolerability as measured by Injection Site reactions
Safety Variable - Immunogenicity as measured by presence of Anti Drug Antibodies | Day 1 of each study period & Day 22 of each study period
  Immunogenicity as measured by presence of Anti Drug Antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Later on management will decide whether to share the data or not